CLINICAL TRIAL: NCT06775730
Title: A Phase 1 Drug-Drug Interaction Study of S-217622 With Combined Oral Contraceptives in Healthy Adult Female Participants
Brief Title: A Drug-Drug Interaction Study of S-217622 With Combined Oral Contraceptives in Healthy Adult Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2403T1219
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Adult Female Participants
MeSH Terms: interventions — ensitrelvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ensitrelvir (Experimental): Participants will receive multiple oral doses of a combined oral contraceptive (COC) (EE and DRSP) once daily for 24 days (Days 1 to 24) (in the fasted state on Days 18 to 24) in the morning. Participants will also receive ensitrelvir high dose on Day 20 and multiple oral doses of ensitrelvir low dose once daily on Days 21 to 24 in the fasted state.
  Interventions: Drug: Ensitrelvir

INTERVENTIONS:
Drug: Ensitrelvir — Ensitrelvir will be administered per schedule specified in the arm description.
  Other Names: S-217622

SUMMARY:
The purpose of this study is to examine the potential for drug-drug interactions.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) within the range of ≥18.5 to ≤30.0 kilograms (kg)/square meter (m^2) at the screening.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and either of the following conditions applies:

  * Is a woman of childbearing potential (WOCBP), having not received any oral contraceptives for at least 28 days prior to the first dose of study intervention, and using a contraceptive method that is highly effective during the treatment period and for at least 14 days after the last dose of study intervention.
  * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.

Key Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Presence (suspected) or history of having breast cancer, endometrial cancer, or cervical cancer.
* Presence of unexplained genital bleeding.
* Participants who have taken injectable or implantable contraceptives, hormonal intrauterine devices, intrauterine hormone-releasing system within 12 months prior to the first dose of study intervention or hormonal contraceptives (intravaginal or transdermal) for 3 months prior to the first dose of study intervention.
* Participants who are otherwise considered ineligible for the study by the investigator for any other reason.

NOTE: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Ethinyl Estradiol (EE) | Predose and up to 24 hours postdose on Days 19, 20, and 24
Cmax of Drospirenone (DRSP) | Predose and up to 24 hours postdose on Days 19, 20, and 24
Time to Reach Cmax (Tmax) of EE | Predose and up to 24 hours postdose on Days 19, 20, and 24
Tmax of DRSP | Predose and up to 24 hours postdose on Days 19, 20, and 24
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUC0-τ) of EE | Predose and up to 24 hours postdose on Days 19, 20, and 24
AUC0-τ of DRSP | Predose and up to 24 hours postdose on Days 19, 20, and 24

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Day 1 up to Day 32
Cmax of Ensitrelvir | Predose and up to 24 hours postdose on Days 20 and 24
Tmax of Ensitrelvir | Predose and up to 24 hours postdose on Days 20 and 24
AUC0-τ of Ensitrelvir | Predose and up to 24 hours postdose on Days 20 and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Early Phase Clinical Unit Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No